CLINICAL TRIAL: NCT00117767
Title: Efficacy and Safety of Terbinafine Compared to Griseofulvin in Children With Tinea Capitis
Brief Title: Terbinafine Compared to Griseofulvin in Children With Tinea Capitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CSFO327C2301
Record Dates: First submitted 2005-06-30; First posted 2005-07-08 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Tinea Capitis
Keywords: Terbinafine, Tinea capitis, pediatric, antifungal
MeSH Terms: conditions — Tinea Capitis | interventions — Terbinafine; Griseofulvin

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- 1 (Experimental): Terbinafine
  Interventions: Drug: Terbinafine hydrochloride (HCl)
- 2 (Active Comparator): Griseofulvin
  Interventions: Drug: Griseofulvin

INTERVENTIONS:
Drug: Terbinafine hydrochloride (HCl) — Terbinafine hydrochloride (HCl) pediatric formulation (minitablets)o.d. administration
  Other Names: Lamisil
  Arms: 1
Drug: Griseofulvin — Griseofulvin pediatric suspension o.d. administration
  Other Names: Grilfulvin V
  Arms: 2

SUMMARY:
Tinea capitis is a dermatophyte infection of the scalp hair follicles, which occurs primarily in children. Hair loss, hair breakage, scaling, plus various degrees of erythema, pustules and pruritus are the primary clinical signs which can be associated with tinea capitis. The infection is caused by a relatively small group of dermatophytes in the genera Trichophyton and Microsporum.

Terbinafine hydrochloride is a synthetic allylamine derivative antifungal agent. This study will evaluate the efficacy and safety of terbinafine in children with tinea capitis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical diagnosis of tinea capitis confirmed by positive KOH determined by the central mycology laboratory.
* Male or female patients who are at least 4 years old and no more than 12 years old.

Exclusion Criteria:

* Patients having a medical condition that alters the absorption and/or metabolism of terbinafine (e.g. liver, renal disease etc.)
* Patients receiving medication that may interfere with the evaluation of the drug's effect
* Patients who have kerions requiring immediate treatment or treatment with systemic corticosteroids and/or systemic antibiotics
* Patients with a history of liver disease or current/active liver disease or with elevation of livery enzymes outside of the normal range corresponding to their age
* Patients who have received recent systemic or topical treatment for tinea capitis within the specified time periods (e.g. systemic antifungals within 2 months of screening visit, topical treatments [e.g. antifungals, corticosteroid preparations, zinc pyrithione or selenium sulfide or tar containing products] within 1 week of screening).
* Patients with a history of systemic lupus erythematosus

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 720
Dates: Start 2004-06; Primary Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Complete cure (negative mycology and clinical cure) rate at Week 10

SECONDARY OUTCOMES:
Clinical cure rate at Week 10
Mycological cure rate at Week 10
Safety of terbinafine

CONTACTS AND LOCATIONS:
Locations (1):
- Novartis Pharmaceuticals, East Hanover, New Jersey, United States

REFERENCES:
- [Background] Elewski BE, Caceres HW, DeLeon L, El Shimy S, Hunter JA, Korotkiy N, Rachesky IJ, Sanchez-Bal V, Todd G, Wraith L, Cai B, Tavakkol A, Bakshi R, Nyirady J, Friedlander SF. Terbinafine hydrochloride oral granules versus oral griseofulvin suspension in children with tinea capitis: results of two randomized, investigator-blinded, multicenter, international, controlled trials. J Am Acad Dermatol. 2008 Jul;59(1):41-54. doi: 10.1016/j.jaad.2008.02.019. Epub 2008 Apr 18. PMID 18378354